CLINICAL TRIAL: NCT06957197
Title: Clinical Comparison of Xenograft With Hydrogel Versus Xenograft Alone in the Socket Preservation After Tooth Extraction: A Randomized Controlled Clinical Trial
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Eslam Mohamed Abdel-monaem, Clinical Comparison of xenograft with hydrogel versus xenograft alone in the socket preservation After tooth extraction: A Randomized controlled Clinical Trial, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Hydrogel in SocketPreservation
Record Dates: First submitted 2025-04-26; First posted 2025-05-04 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-04

CONDITIONS: Socket Perservation
MeSH Terms: interventions — Hydrogels; Transplantation, Heterologous

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial Parallel group study: each group of patients receives a single treatment simultaneously Two arm, superiority trial with allocation ratio 1:1 Positive controlled: both groups receiving treatment. The trial will be carried out by research in OMFS department at faculty of dentistry Cairo University
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention (Experimental): socket preservation via hydrogel + xenograft
  Interventions: Drug: Hydrogel with xenograft
- control (Active Comparator): socket preservation via xenograft alone
  Interventions: Drug: Xenograft

INTERVENTIONS:
Drug: Hydrogel with xenograft — vehicle to hold xenograft
  Arms: intervention
Drug: Xenograft — to maintain the socket
  Arms: control

SUMMARY:
Clinical Comparison of xenograft with hydrogel versus xenograft alone in the socket preservation After tooth extraction: A Randomized controlled Clinical Trial The ideal scaffolds used for alveolar ridge preservation are supposed to show good biocompatibility, mechanical properties, and formability for irregularly shaped bone defects, as well as degradation rates matching bone growth . One of the most used synthetic scaffolds is hydrogel. Hydrogels owning three-dimensional cross-linked network structures have physical and chemical properties like human tissues . They can not only simulate the extracellular matrix (ECM) of bone but also allow the storage, and transport of various growth factors, cytokines, and nutrients due to their high permeability .

DETAILED DESCRIPTION:
Research question:

Is xenograft with hydrogel more effective than xenograft in the socket preservation After tooth extraction? Statement of the problem Alveolar socket preservation therapies aim to maintaining the hard and soft tissue dimensions of the alveolar ridge that are partially lost after tooth extraction as part of the natural physiological healing process. The reduction of alveolar bone volume following tooth extraction may interfere with placement of implants and affect the treatment and success of fixed or removable prosthesis with regard to function and esthetics. Alveolar socket preservation via socket filling with a bone graft can be an effective therapy to prevent physiologic bone loss after extraction of teeth in both the horizontal and the vertical dimension - Rationale for conducting a study The ideal scaffolds used for alveolar ridge preservation are supposed to show good biocompatibility, mechanical properties, and formability for irregularly shaped bone defects, as well as degradation rates matching bone growth . One of the most used synthetic scaffolds is hydrogel. Hydrogels owning three-dimensional cross-linked network structures have physical and chemical properties like human tissues . They can not only simulate the extracellular matrix (ECM) of bone but also allow the storage, and transport of various growth factors, cytokines, and nutrients due to their high permeability .

Explanation for choice of comparators:

The comparator here is the well-known technique of extraction socket preservation with xenograft ,as preservation of extraction sockets has become a more popular treatment over the last 15 years, Xenografts are the most commonly used in regenerative therapy for alveolar ridge preservation as they contain similar hydroxyapatite content to that of natural bone which allows the graft to revascularize and be replaced by new bone, also the intervention and comparator have a common feature of being enhance bone formation by promoting osteoconduction, osteoinduction, and osteogenesis.

III. Methods A) Participants, interventions & outcomes 9. Study settings: This study will be conducted on number cases of sockets need to be preserved, (10) cases with xenograft alone and (10) cases with xenograft with hydrogel selected from the outpatient clinic, OMFS departments at Faculty of Dentistry - Cairo University.

10. Eligibility criteria: Inclusion criteria: Adult, systemically healthy patients with hopeless infected teeth and nonrestorable remaining structure or root.

Exclusion criteria: Systemic or local disease/ condition that would compromise post-operative healing (e.g. Diabetics, patients who in need for systemic corticosteroids).

11. Interventions:

I. Pre-Surgical Preparation:

1. clinical examination: History data will be gathered including personal data, medical and surgical history, and familial history.
2. all patients will be submitted to full mouth supragingival and subgingival scaling and root planning (SRP) procedures prior to extraction.
3. radiographic examination: cbct for all patients.

   II. Surgical Procedure:

   -After local anesthesia , A forceps of anatomic design and periotome will be used to retrieve the tooth from the alveolus.
   * Curettage of the socket will be followed by irrigation with 0.9 saline concentration.
   * Then the socket will be filled with graft materials according to group types. Only xenograft in group I, xenograft mixed with hydrogel in group II,

     -.A gelfoam is trimmed to completely cover the socket.
   * Figure 8 sutures will be done to achieve primary closure of the surgical wound.

   Post-operative care:

   -All the patients will be instructed to refrain from interfering with the wound or sutures, or using tooth brushing in the operated area.

   -Medications (Augmentin1gm tablet (875mg Amoxicillin and potassium clavulanate equivalent to 125mg of clavulanic acid) will be prescribed twice daily for 5days ,Cataflam 50mg tablet will be prescribed twice daily for 5 days to minimize the postoperative pain.A 0.2% chlorhexidine digluconate Hexitol twice daily for the first two postoperative weeks will be also recommended.

   12. Outcomes:

   Primary outcome:

   quantity of bone (bone height): measured radiographically

   Secondary outcome:
   1. quantity of bone (bone width): measured radiographically
   2. quality of bone (area percentage pf newly formed bone after 3 months) this outcome will be measured by histomorphometric analysis by core biopsy
   3. other complication: pain, edema, infection, fistula development or dehiscence by clinical examination in follow up visits

   Prioritization of Outcome Outcome Method of Measurement Unit of Measurement Primary outcome Quantity of bone (bone height) Radiographically mm Secondary outcome Quantity of bone (bone width) Radiographically mm Quality of bone Histomorphometric analysis by core biopsy Area percentage of newly formed bone
   * Pain
   * Edema
   * Infection
   * Fistula development -visual analogue scale
   * linear measurement
   * clinically
   * clinically -numbers
   * mm
   * yes or no
   * yes or no

     13. Participant timeline:

   Study steps Enrollment Post-allocation Day Of Surgery Follow-up Time point T0 T1 T2 T3 T4 Enrollment Eligibility screening ✓ Informed consent ✓ Pre-operative Documentation and CBCT ✓ Intervention Surgical procedure ✓ Postoperative Core Biopsy and CBCT ✓

   T1: Intra-operative T2: 3 days post-operative T3: 1-week post-operative T4: 3 months post-operative

   14. Sample size: A total of (22) cases. i.e. (11) cases per group In a previous study by Shokry et al in 2023 the alveolar bone height using xenograft after 3 months showed a standard deviation of 0.4. If the true difference in the experimental and control means is 0.5 we will need to study 11 patients per group to be able to reject the null hypothesis that the population means of the experimental and control groups are equal with probability (power) 0.8. The Type I error probability associated with this test of this null hypothesis is 0.05. Sample size was increased by 15% to compensate for possible dropouts to reach 13 patients per group. Sample size was calculated using PS Power and Sample for windows version 3.1.6 using independent t test.

   15. Recruitment: Patients will be selected by the supervisors and the researchers from outpatient clinic of OMFS departments at Faculty of Dentistry - Cairo University will start in December 2024. Screening of patients according to the inclusion and exclusion criteria and will continue until the target population is achieved. Identifying and recruiting potential subjects is achieved through patient database.

   B) Assignment of interventions 16. Allocation: 16a. Randomization: The total sample size (n=) and the sample sizes in each group are pre-specified exactly and are under the direct control of the investigator. 1- Method of random sequence generation: (computerized random number generator). 2- Allocation ratio: (1:1). 3- Type of randomization: simple 16b. Allocation concealment mechanism: The cards will take the generated sequence numbers one number for each card then these cards will be placed within opaque sealed envelopes. Then these Envelops will be placed in a container (box), each participant will grasp one envelop blindly during the preoperative preparation 16c. Implementation Author is the person who will generate the allocation sequence. Principal investigator will enroll the participants and assign the participants for intervention.

   17. Masking/blinding: the interventions used in this trial are easily blinded by the participants and the investigator, and statistician will be blinded

   C) Data collection, management, and analysis:

   18. Data collection methods: Author who will be responsible for outcomes assessment. Information on demographic data and past and concurrent medical history will be obtained by interviewing the patient. During (pre-operative visit); Data regarding personal information, medical history and familial history will be obtained. At (operative procedure (including surgical procedure- intraoperative complications- operation time) and postoperative complication will be recorded each in the specified section in prepared form. In each follow-up visit symptoms, clinical features,

   - For outcome evaluation and instruments used : follow-up intervals will be 3 days, 1 week, 3 months, clinical and radiographic. Plans to promote participant retention & complete follow-up: Telephone numbers and address of the patient included in the study will be recorded. All patients will be given a phone call and text message before the next appointment.

   19. Data management: All data will be entered electronically. Patient files are to be stored in numerical order and stored in a secure and accessible place. All data will be maintained in storage for 1 year after completion of the study.

   20. Statistical methods:

a. Outcome: A suitable statistical test will be used for one group. b. Methods for any Additional Analysis: No additional subgroup analysis.

Statistical analysis:

Data will be analyzed using Medcalc software, version 22 for windows (MedCalc Software Ltd, Ostend, Belgium). Continuous data will be described using mean and standard deviation. Intergroup comparison will be performed using independent t test and intragroup comparison will be done using repeated measures ANOVA followed by tukey post hoc test. Categorical data will be described as frequency and percentage. Intergroup comparisons between categorical variables will be performed using the chi square test, while intragroup comparisons within each intervention will be performed using Cochran's Q test followed by pairwise multiple comparisons. A p-value less than or equal to 0.05 will be considered statistically significant and all tests will be two tailed. Statistical power of the study will be set at 80 % with 95 % confidence level.

D) Data monitoring:

21. Monitoring In most protocols, no formal data monitoring committee will be needed since most of studies in Faculty of Dentistry are with known minimal risks.

22. Harms

Intra-operative complications:

* Bleeding: avoided by -Proper hemostatic measure

Post-operative complications:

* Infection & wound dehiscence: avoided by 1-Appropriate antibiotic. 2- Strict wound hygiene measures 23. Audit Auditing of the study design will be done by the evidence-based committee - Faculty of Dentistry - Cairo University

ELIGIBILITY:
Inclusion Criteria:

* Adult, systemically healthy patients with hopeless infected teeth and nonrestorable remaining structure or root.

Exclusion Criteria:

* Systemic or local disease/ condition that would compromise post-operative healing (e.g. Diabetics, patients who in need for systemic corticosteroids).

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 26 (Estimated)
Dates: Start 2025-09-22 (Estimated); Primary Completion 2026-07-20 (Estimated); Study Completion 2026-08-20 (Estimated)

PRIMARY OUTCOMES:
Quantity of bone (bone height) | 3 mounths
  Method of Measurement ;Radiographically Unit of Measurement ;mm

SECONDARY OUTCOMES:
Quantity of bone (bone width) | 3 mounths
  Method of Measurement Radiographically Unit of Measurement mm
Quality of bone | 3 mounths
  Method of Measurement Histomorphometric analysis by core biopsy Unit of Measurement Area percentage of newly formed bone
Pain value | 1 week
  Method of Measurement visual analogue scale Unit of Measurement numbers
Infection | 1 week
  Method of Measurement clinically Unit of Measurement yes or no
Edema | 1 week
  Method of Measurement
  -linear measurement Unit of Measurement mm
Fistula development | 1 week
  Method of Measurement clinically Unit of Measurement
  -yes or no

CONTACTS AND LOCATIONS:
Overall Officials: socket preservation, Study Director — Cairo University
Locations (1):
- Cairo University, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No